CLINICAL TRIAL: NCT02506907
Title: Vanderbilt Assessment of Multi-modal MRI in Patients At-Risk for Stroke With Intracranial Stenosis
Brief Title: Characterizing Hemodynamic Compensation in Patients With Intracranial Stenosis
Acronym: VAMMPRIS
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Manus Donahue, Associate Professor of Radiology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: VUMC-VAMMPRIS
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Stroke; Intracranial Stenosis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atherosclerotic: Patients with atherosclerotic intracranial stenosis

SUMMARY:
The overall aim of this work is to assess the relationship between stroke risk and hemodynamic compensation strategies, as measured using a novel 3.0 Tesla MRI protocol, in patients with symptomatic intracranial (IC) steno-occlusive disease. Recent studies have shown high two-year ischemic stroke rates in symptomatic patients with IC arterial stenosis. Therapy for IC stenosis patients includes revascularization with angioplasty, IC stenting, or bypass, however identification of patients most likely to benefit from these more aggressive interventions, rather than medical management alone, has been problematic. Accurate measurements of hemodynamic compromise are likely required to better define stroke risk and guide treatment decisions. Specifically, in IC stenosis patients with compromised cerebral perfusion pressure (CPP), the extent of hemodynamic compromise reflects the autoregulatory capacity of vasculature to increase arterial cerebral blood volume (aCBV) and/or develop collaterals to supplement cerebral blood flow (CBF). The prevalence of CBF collateralization and aCBV autoregulation has been hypothesized to correlate uniquely with stroke risk, however the extent of this correlation has been debated. The critical barrier to stratifying stroke risk rests with a lack of (i) methodology for measuring multiple hemodynamic factors with high specificity and (ii) noninvasive approaches capable of monitoring longitudinal progression of impairment. The investigators have demonstrated the clinical utility of relatively new, noninvasive MRI approaches for assessing cerebrovascular reactivity (CVR), aCBV, and collateral CBF. The investigators hypothesize that stroke risk can be more completely evinced from collective measurements of these parameters. Therefore, the investigators propose to implement a novel, validated hemodynamic MRI protocol to assess tissue-level impairment and compensation strategies in patients with IC stenosis. Using a collective approach combining measurements of collateral CBF, aCBV and CVR in multiple brain regions, in conjunction with a statistical model incorporating the above variables as possible prognostic factors, the investigators will quantify the extent to which two-year stroke risk is associated with hemodynamic compensation mechanisms. The noninvasive and multi-faceted scope of this investigation is intended to expand the diagnostic stroke infrastructure and elucidate new hemodynamic prognostic indicators of stroke in this high-risk population.

DETAILED DESCRIPTION:
The overall aim of this work is to assess the relationship between stroke risk and hemodynamic compensation strategies, as measured using a novel 3.0 Tesla (T) MRI protocol, in patients with symptomatic intracranial (IC) steno-occlusive disease. Recent studies have shown high two-year ischemic stroke rates of approximately 20% in symptomatic IC stenosis patients. Aggressive therapy for IC stenosis patients includes revascularization with angioplasty, IC stenting, or bypass, however identification of patients most likely to benefit from these more aggressive interventions, rather than medical management alone, has been problematic. Accurate measurements of hemodynamic compromise are likely required to better define stroke risk and guide treatment decisions. Specifically, in IC stenosis patients with compromised cerebral perfusion pressure (CPP), the extent of hemodynamic compromise reflects the autoregulatory capacity of vasculature to increase arterial cerebral blood volume (aCBV) and/or develop collaterals to supplement cerebral blood flow (CBF). The prevalence of CBF collateralization and aCBV autoregulation has been hypothesized to correlate uniquely with stroke risk, however the extent of this correlation is debated.

The critical barrier to stratifying stroke risk rests with a lack of (i) methodology for measuring multiple hemodynamic factors with high specificity and (ii) noninvasive approaches capable of monitoring longitudinal progression of impairment. The investigators have demonstrated the clinical utility of relatively new, noninvasive MRI approaches for assessing cerebrovascular reactivity (CVR), aCBV, and collateral CBF. These approaches have been optimized and feasibility assessed in healthy volunteers or isolated clinical studies, however comparatively little information is available regarding the relationship between these collective measures and stroke risk. Therefore, the investigators propose to complement established angiographic and structural imaging with more novel, validated hemodynamic measurements to assess tissue-level impairment and compensation strategies in patients with IC stenosis. Using a collective approach combining measurements of collateral CBF, aCBV and CVR in multiple brain regions, in conjunction with a statistical model incorporating the above parameters as possible prognostic factors, the investigators will quantify the extent to which two-year stroke risk is associated with hemodynamic compensation mechanisms in a population of symptomatic IC stenosis patients. The noninvasive and multi-faceted scope of this investigation is intended to expand the diagnostic stroke infrastructure and elucidate new hemodynamic prognostic indicators of stroke in this high-risk population.

Hypothesis (1). Changes in collateral CBF with hypercarbic stimulation positively correlate with two-year stroke incidence in symptomatic IC stenosis patients.

Aim (1). By separately magnetically labeling blood water in different feeding arteries (8), the investigators will use a tested vessel-selective arterial spin labeling (VS-ASL) approach and a calculated perfusion asymmetry index to noninvasively assess changes in collateral CBF patterns in patients with IC stenosis. IC stenosis (n=90) patients will be monitored for two years during which their known stroke incidence is 20%. Stroke incidence will be recorded and separate correlations between perfusion asymmetry and stroke risk will be assessed.

Hypothesis (2). Regionally reduced CVR, indicative of vascular steal phenomena, and elevated aCBV, will positively correlate with two-year stroke incidence in symptomatic IC stenosis patients.

Aim (2). CVR, as measured using the blood oxygenation level-dependent (BOLD) MRI signal change in response to hypercarbia, will be used to assess cerebrovascular reserve. The inflow vascular-space-occupancy with dynamic subtraction (iVASO-DS) approach, which we have developed and demonstrated in patients, will be applied to assess baseline aCBV. For the same patients as in Aim 1, CVR dynamics and aCBV will be statistically assessed for unique relationships with two-year stroke incidence.

Hypothesis (3). Collateral CBF, autoregulatory aCBV, and CVR will correlate unequally with two-year stroke incidence, the extent of which can be quantified using a multi-component prediction model.

Aim (3). The investigators will build a statistical prediction model, using collateral CBF, aCBV and CVR as prognostic factors, to quantify the extent to which trends in the above parameters collectively contribute to stroke risk. The high two-year stroke rate (20%) and large number of admitted patients with symptomatic IC stenosis, will enable this study to detect hypothesized group differences with high statistical power.

This work is an extension of recent methodological work whereby a novel, collective compensatory hemodynamic protocol is applied to a specific clinical population to understand prognostic potential. Successful completion should provide new information on tissue hemodynamics and stroke risk in patients that can be used to guide management decisions, ultimately reducing stroke incidence in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age 18-85, inclusive)
2. Symptomatic (TIA or ischemic stroke) in the hemispheric carotid territory of vascular stenosis
3. Vascular imaging demonstrating large vessel IC stenosis>50% or occlusion of IC carotid or MCA
4. Sub-acute stroke patients who have received intravenous or intra-arterial treatments
5. Sub-acute stroke patients ineligible for conventional acute stroke intervention. Language comprehension intact, motor aphasia mild or absent, competent to give informed consent
6. Most recent qualifying TIA or stroke within 60 days prior to performance date of hemodynamic MRI

Exclusion Criteria:

1. ECA stenosis > 70% determined by MRA, CTA, or DSA.
2. Acute stroke patients presenting with anterior circulation stroke onset eligible for intervention with intra-arterial thrombolysis or mechanical thrombectomy
3. MRI contraindications (e.g. non-compatible implants, pregnancy, etc.)
4. Non-atherosclerotic cervical or intracranial stenosis
5. Heart disease likely to cause cerebral ischemia, including cardiomyopathy with ejection fraction<25%, prosthetic valve, infective endocarditis, sick sinus syndrome, myxoma, left atrial or ventricular thrombus
6. Existing condition likely to lead to death within 2 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial stenosis who have had a stroke within the past 60 days
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06-06 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Stroke | Two years
  An overt or silent stroke (on MRI) in two years

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States